CLINICAL TRIAL: NCT06237517
Title: Assessment of Vasomotion of People With Idiopathic Chilblains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Petros Dinas, Senior Researcher in human physiology, University of Thessaly, University of Thessaly
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1888
Record Dates: First submitted 2024-01-21; First posted 2024-02-01 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Chilblains; Perniosis; Thermoregulation
Keywords: Non-freezing cold injuries; Chilblains; Perniosis; Skin lesions; Vasomotion
MeSH Terms: conditions — Chilblains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Progressive acclimation of healthy individuals with Idiopathic Chilblains (Experimental): Throughout the experiment, the participants remained seated in a sitting position. The trial began with the chamber's temperature at 22-24°C and 40-50% (relative humidity) for 20 minutes. After this period, the temperature within the chamber dropped by 4 degrees every 20 minutes. After 80 minutes, the temperature was maintained at 10°C and 40-50% (relative humidity) for 15 minutes, and an occlusion foot test for 15 minutes, and an occlusion foot test (5 minutes ''baseline'' phase, 5 minutes ''occlusion'' phase, and 5 minutes ''release'' phase) was performed to observe any hemodynamic changes in the foot. Participants provided blood and urine samples before and following the trial.
  Interventions: Behavioral: Assessment of Vasomotion of People With Idiopathic Chilblains
- Progressive acclimation of healthy individuals with Idiopathic Chilblains (Rewarming Phase) (Experimental): Throughout the experiment, the participants remained seated in a sitting position. The trial began with the chamber's temperature at 22-24 °C and 40-50% relative humidity for 20 minutes. After this period, the temperature within the chamber dropped by 4 degrees every 20 minutes. After 80 minutes (the chamber's temperature was 10°C and 40-50%), a radiator heater was placed in front of the participants to increase the temperature of their extremities. Simultaneously, the investigators increased the temperature of the chamber to 22-24 °C and 40-55% relative humidity, and the participants remained in the same sitting position for 20 minutes. Following this period, an occlusion foot test was performed to observe any hemodynamic changes in the foot. The test consisted of a 5-minute ''baseline'' phase, a 5-minute ''occlusion'' phase, and a 5-minute ''release'' phase. Before and after the trial, participants provided blood and urine samples.
  Interventions: Behavioral: Assessment of Vasomotion of People With Idiopathic Chilblains
- Progressive acclimation of healthy individuals without Idiopathic Chilblains (Active Comparator): Throughout the experiment, the participants remained seated in a sitting position. The trial began with the chamber's temperature at 22-24°C and 40-50% (relative humidity) for 20 minutes. After this period, the temperature within the chamber dropped by 4 degrees every 20 minutes. After 80 minutes, the temperature was maintained at 10°C and 40-50% (relative humidity) for 15 minutes, and an occlusion foot test for 15 minutes, and an occlusion foot test (5 minutes ''baseline'' phase, 5 minutes ''occlusion'' phase, and 5 minutes ''release'' phase) was performed to observe any hemodynamic changes in the foot. Participants provided blood and urine samples before and following the trial.
  Interventions: Behavioral: Assessment of Vasomotion of People With Idiopathic Chilblains
- Progressive acclimation of healthy individuals without Idiopathic Chilblains (Rewarming Phase) (Active Comparator): Throughout the experiment, the participants remained seated in a sitting position. The trial began with the chamber's temperature at 22-24 °C and 40-50% relative humidity for 20 minutes. After this period, the temperature within the chamber dropped by 4 degrees every 20 minutes. After 80 minutes (the chamber's temperature was 10°C and 40-50%), a radiator heater was placed placed in front of the participants to raise the temperature of their extremities. Simultaneously, the investigators increased the chamber temperature to 22-24 °C and 40-55% relative humidity, and the participants remained in the same sitting position for 20 minutes. Following this period, an occlusion foot test was performed to observe any hemodynamic changes in the foot. The test consisted of a 5-minute ''baseline'' phase, a 5-minute ''occlusion'' phase, and a 5-minute ''release'' phase. Before and after the trial, participants provided blood and urine samples.
  Interventions: Behavioral: Assessment of Vasomotion of People With Idiopathic Chilblains
- Thermoneutral environment healthy participants with Idiopathic Chilblains (Baseline) (Experimental): Throughout the experiment, the participants remained seated in a sitting position. The trial began with the chamber's temperature at 22-24°C and 40-50% (relative humidity) for 20 minutes. After 20 minutes, the temperature was maintained at 22°C and 40-50% (relative humidity) for 15 minutes, and an occlusion foot test was conducted (5 minutes ''baseline'' phase, 5 minutes ''occlusion'' phase, and 5 minutes ''release'' phase), to observe any hemodynamic changes in the foot.
  Interventions: Behavioral: Assessment of Vasomotion of People With Idiopathic Chilblains
- Thermoneutral environment healthy participants without Idiopathic Chilblains (Baseline) (Active Comparator): Throughout the experiment, the participants remained seated in a sitting position. The trial began with the chamber's temperature at 22-24°C and 40-50% (relative humidity) for 20 minutes. After 20 minutes, the temperature was maintained at 22°C and 40-50% (relative humidity) for 15 minutes, and an occlusion foot test was conducted (5 minutes ''baseline'' phase, 5 minutes ''occlusion'' phase and 5 minutes ''release'' phase), to observe any hemodynamic changes in the foot.
  Interventions: Behavioral: Assessment of Vasomotion of People With Idiopathic Chilblains

INTERVENTIONS:
Behavioral: Assessment of Vasomotion of People With Idiopathic Chilblains — Investigation of vasomotion of people with and without idiopathic chilblains

SUMMARY:
Chilblains, also known as perniosis, is a non-freezing cold injury causing painful inflammatory skin lesions. Chilblains typically affect the dorsal feet or hands, causing inflammatory skin lesions that are often painful, and their pathogenesis remains only partly understood. To improve diagnosis and management, it is vital to focus entirely on chilblains and consider the patient-related and environmental factors that characterize this disorder. Because of this, it's critical to investigate the thermoregulatory function, of individuals with idiopathic chilblains while they are exposed to various environmental conditions (cold and neutral environments).

DETAILED DESCRIPTION:
The participants will visit the laboratory three times. The environmental scenarios were randomly allocated for each participant.

The three different environments will be as follows:

1. Thermoneutral environment 22-24°C and 40-50% relative humidity for 15 minutes.
2. Thermoneutral environment of 22-24°C and 40-50% relative humidity, the temperature within the chamber was decreased by 4 degrees every 20 minutes.
3. Thermoneutral environment of 22-24°C and 40-50% relative humidity, the temperature within the chamber was decreased by 4 degrees every 20 minutes. After 80 minutes (the chamber's temperature will be 10°C and 40-50% relative humidity), the investigators increased the chamber temperature to 22-24 °C and 40-55% relative humidity, and the participants remained in the same sitting position for 20 minutes.

All participants had antinuclear antibodies blood testing for a suspected autoimmune disease such as lupus, rheumatoid arthritis, or scleroderma. Participants were provided blood (C-reactive protein and serum Cortisol) before, immediately after, and 24 hours after each trial and urine samples before and following the trials.

Anthropometric data [self-reported age, self-reported body stature, and body mass (DXA, Lunar, GE Healthcare Boston, Massachusetts, U.S.)] will be collected at the beginning of the first visit. Investigators recorded the medical history of all the participants. During the study, continuous heart rate and heart rate variability (Polar Team2. Polar Electro Oy, Kempele, Finland), core temperature (telemetric capsules BodyCap, Caen, France), mean skin temperature (wireless thermistors iButtons type DS1921H, Maxim/Dallas Semiconductor Corp., USA), finger temperature, skin blood flow (laser Doppler flow-meter PeriFlux System 5010, Stockholm, Sweden), and tissue oxygenation changes (Near-Infrared Spectroscopy, PortaLite mini, Artinis Medical Systems, Zetten, Netherlands) will be collected. Skin temperature data collected from seven sites (forehead, arm, thigh, hand, foot, tibialis anterior, navel) and will be expressed as mean skin temperature according to the formula of Hardy/Bubois (Tsk = [0.7 (forehead) + 0.14 (arm) + 0.05 (hand) + 0.07 (foot) + 0.13 (tibialis anterior) + 0.19 (thigh) + 0.35 (navel)]. Hydration status was assessed using a handheld refractometer (ATAGO Ltd, Tokyo, Japan) and determined as either euhydrated (USG < 1.020) or dehydrated (USG ≥ 1.020) according to the current guidelines. Questionnaires (thermal sensation scale: -3 = cold; +3 = hot) assessed participants' thermal comfort/sensation and pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals with and without idiopathic chilblains.

Exclusion Criteria:

* Non-healthy individuals or any underlying connective tissue disorders (particularly: Raynaud syndrome/phenomenon, Systemic Lupus Erythematosus, Scleroderma)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Heart rate | 1 hour and 35 minutes (trial without rewarming), 1 hour and 55 minutes (trial with rewarming)
  Heart rate were continuously monitored using a Polar Team system (Polar® Team 2, Polar Electro Oy, Kempele, Finland
Heart rate variability | 1 hour and 35 minutes (trial without rewarming), 1 hour and 55 minutes (trial with rewarming)
  Heart rate variability were continuously monitored using a Polar Team system (Polar® Team 2, Polar Electro Oy, Kempele, Finland
Skin blood flow | 1 hour and 35 minutes (trial without rewarming), 1 hour and 55 minutes (trial with rewarming)
  Skin blood flow was measured throughout the entire protocol with a laser Doppler flowmeter ((PeriFlux System 5010, function unit; Perimed, Stockholm, Sweden, PeriFlux 4000, Perimed, Stockholm, Sweden) at right and left index finger and right and left index toe.
Skin temperature | 1 hour and 35 minutes (trial without rewarming), 1 hour and 55 minutes (trial with rewarming)
  Skin temperature (forehead, arm, thigh, hand, foot, tibialis anterior, navel) was continuously monitored using iButton sensors type DS1921 H, Maxim/Dallas Semiconductor Corp., USA.
Finger temperature | 1 hour and 35 minutes (trial without rewarming), 1 hour and 55 minutes (trial with rewarming)
  Finger temperature were monitored throughout the trial using a data logger interfacing with a computer to allow for their continuous monitoring by the investigators.
Hemoglobin oxygen saturation in a localized tissue (foot) | 1 hour and 35 minutes (trial without rewarming), 1 hour and 55 minutes (trial with rewarming)
  Hemoglobin oxygen saturation in a localized tissue were monitored throughout the trial at 10Hz and data duration 919.2s using (Near-Infrared Spectroscopy, PortaLite mini, Artinis Medical Systems, Zetten, Netherlands).
Body core temperature | 1 hour and 35 minutes (trial without rewarming), 1 hour and 55 minutes (trial with rewarming)
  Core body temperature was assessed using telemetric capsules (e-Celsius, BodyCap, Caen, France) which were ingested by the participants 2 hours before of each trial.
Thermal comfort | Change from baseline thermal comfort at 20th, 40th, 60th, and 80th minute (for trial without warming - 1 hour and 35 minutes), and at 20th, 40th, 60th, 80th, and 100th minute (for trial with warming - 1 hour and 55 minutes)
  Thermal comfort was assessed via the thermal comfort scale (1 = comfortable; 5 = extremely uncomfortable).
Thermal sensation | Change from baseline thermal sensation at 20th, 40th, 60th, and 80th minute (for trial without warming - 1 hour and 35 minutes), and at 20th, 40th, 60th, 80th, and 100th minute (for trial with warming - 1 hour and 55 minutes)
  Thermal sensation was assessed via the thermal sensation scale (-3 = cold; +3 = hot)
Blood samples | Participants were given blood samples at baseline, at 1 hour and 35 minutes (trial without rewarming)/1 hour and 55 minutes (trial with rewarming), and 24 hours after each trial.
  Participants were provided blood samples (C-reactive protein and Cortisol).
Urine sample | Participants were given urine samples at baseline, at 1 hour and 35 minutes (trial without rewarming)/1 hour and 55 minutes (trial with rewarming), and 24 hours after each trial.
  Participants were provided urine samples (urine specific gravity)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Flouris, PhD, Principal Investigator — FAME Lab, Department of Exercise Science, University of Thessaly Tríkala, Thessaly, Greece, 42100
Locations (1):
- FAME Lab, Department of Exercise Science, University of Thessaly Tríkala, Thessaly, Greece, 42100, Trikala, Greece